CLINICAL TRIAL: NCT06338735
Title: Ultra-High Frequency Ultrasonography (UHFUS) Evaluation of Salivary Glands in Patients With Suspected Sjögren's Syndrome
Brief Title: Ultra-High Frequency Ultrasonography in Sjögren's Syndrome
Acronym: UltraSjögren
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Rossana Izzetti, Researcher at the Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine of the University of Pisa, Principal Investigator, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14540
Record Dates: First submitted 2024-03-21; First posted 2024-04-01 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sjogren's Syndrome
Keywords: ultra-high frequency ultrasonography; diagnostic imaging; Sjogren's syndrome; salivary glands
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sjogren's syndrome (Experimental): patients with Sjogren's syndrome diagnosed according to the ACR/EULAR criteria
  Interventions: Other: Ultra-High Frequency Ultrasound scan of minor salivary glands

INTERVENTIONS:
Other: Ultra-High Frequency Ultrasound scan of minor salivary glands — Patients will undergo ultra-high frequency ultrasonography (70 MHz) of minor salivary glands, and the scans will be assessed using the OMERACT scoring system. Score 0 will be assigned in the presence of normal glandular tissue, Score 1 will correspond to mild glandular alteration, fine echogenicity or diffuse hypo-echogenicity, Score 2 will be assigned to moderate glandular alteration and focal hypoechoic areas with partial conservation of normal parenchyma, while in Score 3 diffuse presence of hypoechoic areas in the absence of normal glandular parenchyma with glandular fibrosis will be observed.

SUMMARY:
Patients diagnosed with a diagnosis of Sjogren's syndrome performed according to the ACR/EULAR criteria will be included in the study. Sjogren's syndrome diagnosis will be performed following a complete diagnostic work-up involving rheumatologic assessment, glandular functional tests, and blood testing for anti-Ro(SSA) antibodies. Conventional ultrasonography of major salivary glands and ultra-high frequency ultrasonography (70 MHz) of minor salivary glands will be performed, and the scans assessed using the Outcome Measures in Rheumatology (OMERACT) scoring system (Score 0 normal glandular tissue, Score 1 mild glandular alteration, fine echogenicity or diffuse hypo-echogenicity, Score 2 moderate glandular alteration and focal hypoechoic areas with partial conservation of normal parenchyma, Score 3 diffuse presence of hypoechoic areas in the absence of normal glandular parenchyma with glandular fibrosis. Focus Score will be assessed following biopsy of minor salivary glands.

DETAILED DESCRIPTION:
Primary Sjögren's syndrome is a complex autoimmune disease involving the exocrine salivary and lachrymal glands, with a progressive functional impairment caused by lymphocytic infiltration in the glandular tissue. The diagnosis is currently performed according to the criteria established in 2016 by the American College of Rheumatologists/European League Against Rheumatism (ACR/EULAR) and relies on 5 items, namely i) histologic Focus Score (FS) ≥1, ii) positivity to Anti-SSA (Ro) antibodies, iii) Ocular staining score ≥ 5 (or van Bijsterfeld score ≥ 4) on at least one eye, iv) Schirmer test ≤ 5 mm/5min on at least one eye and v) Unstimulated Salivary Flow Rate (USFR) ≤ 0.1 ml/min. Focus Score and positivity to antibodies are items with a weight of 3 points each, while the other items are assigned score 1. Diagnosis is performed with a total score ≥ 4 when summing the weights. While the improvement in the sensitivity of ACR/EULAR classification criteria by 5-10% has been previously reported for ultrasonography of major salivary glands, at present no evidence is available for minor salivary glands. Minor salivary glands ultrasonography with the use of ultra-high frequencies up to 70 MHz has been recently introduced in the diagnostic work-up of Sjögren's syndrome, and involves the assessment of glandular ultrasonographic structural alterations through the application of the Outcome Measures in Rheumatology (OMERACT) scoring system, which is routinely used for major salivary glands. The present study therefore aims to assess the correlation between minor salivary glands ultrasonography and ACR/EULAR items, in order to evaluate whether this technique may integrate the current evaluation of Sjögren's syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years of age
* clinical suspect of Sjogren's syndrome
* acceptance to undergo complete Sjogren's Syndrome diagnostic work-up
* acceptance to be included in the study.

Exclusion Criteria:

* pregnancy or breastfeeding
* any acute or chronic condition that would limit the ability of the patient to participate in the study
* refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
OMERACT score | 1 month
  Evaluation of ultrasonographic scans with the Outcome Measures in Rheumatology (OMERACT) scoring system, ranging between Score 0 (normal glandular tissue) and 3 (diffuse presence of hypoechoic areas in the absence of normal glandular parenchyma with glandular fibrosis )
Correspondence between ultrasonography and histology | 1 month
  Evaluation of the concordance between ultrasonographic score of minor salivary glands assessed with Outcome Measures in Rheumatology (OMERACT) scoring system (scores 0-3) and histology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanc N, Jousse-Joulin S, Abacar K, Cimsit C, Cimsit C, D'Agostino MA, Naredo E, Hocevar A, Finzel S, Pineda C, Keen H, Iagnocco A, Hanova P, Schmidt WA, Mumcu G, Terslev L, Bruyn GA. The Novel OMERACT Ultrasound Scoring System for Salivary Gland Changes in Patients With Sjogren Syndrome Is Associated With MRI and Salivary Flow Rates. J Rheumatol. 2024 Mar 1;51(3):263-269. doi: 10.3899/jrheum.2023-0202. PMID 37914219
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome: A Consensus and Data-Driven Methodology Involving Three International Patient Cohorts. Arthritis Rheumatol. 2017 Jan;69(1):35-45. doi: 10.1002/art.39859. Epub 2016 Oct 26. PMID 27785888
- [Background] Brito-Zeron P, Baldini C, Bootsma H, Bowman SJ, Jonsson R, Mariette X, Sivils K, Theander E, Tzioufas A, Ramos-Casals M. Sjogren syndrome. Nat Rev Dis Primers. 2016 Jul 7;2:16047. doi: 10.1038/nrdp.2016.47. PMID 27383445
- [Result] Ferro F, Izzetti R, Vitali S, Aringhieri G, Fonzetti S, Donati V, Dini V, Mosca M, Gabriele M, Caramella D, Baldini C. Ultra-high frequency ultrasonography of labial glands is a highly sensitive tool for the diagnosis of Sjogren's syndrome: a preliminary study. Clin Exp Rheumatol. 2020 Jul-Aug;38 Suppl 126(4):210-215. Epub 2020 Oct 23. PMID 33095145
- [Result] Donati V, Ferro F, Governato G, Fulvio G, Izzetti R, Nardini V, Baldini C. Total area of inflammatory infiltrate and percentage of inflammatory infiltrate identify different clinical-serological subsets of primary Sjogren's syndrome better than traditional histopathological parameters. Clin Exp Rheumatol. 2020 Jul-Aug;38 Suppl 126(4):195-202. Epub 2020 Oct 23. PMID 33095147
- [Result] Izzetti R, Ferro F, Vitali S, Nisi M, Fonzetti S, Oranges T, Donati V, Caramella D, Baldini C, Gabriele M. Ultra-high frequency ultrasonography (UHFUS)-guided minor salivary gland biopsy: A promising procedure to optimize labial salivary gland biopsy in Sjogren's syndrome. J Oral Pathol Med. 2021 May;50(5):485-491. doi: 10.1111/jop.13162. Epub 2021 Feb 15. PMID 33501696
- [Result] Fulvio G, Donati V, Izzetti R, Fonzetti S, La Rocca G, Ferro F, Baldini C. Correspondence between minor salivary glands ultra-high frequency ultrasonography and histology: a case report of severe/atypical lymphoid infiltrate in Sjogren's syndrome. Clin Exp Rheumatol. 2022 Dec;40(12):2474-2475. doi: 10.55563/clinexprheumatol/rdbm3h. Epub 2022 Dec 20. No abstract available. PMID 36541238
- [Result] Fulvio G, Izzetti R, Aringhieri G, Donati V, Ferro F, Gabbriellini G, Mosca M, Baldini C. UHFUS: A Valuable Tool in Evaluating Exocrine Gland Abnormalities in Sjogren's Disease. Diagnostics (Basel). 2023 Aug 26;13(17):2771. doi: 10.3390/diagnostics13172771. PMID 37685309
- [Result] Izzetti R, Fulvio G, Nisi M, Gennai S, Graziani F. Reliability of OMERACT Scoring System in Ultra-High Frequency Ultrasonography of Minor Salivary Glands: Inter-Rater Agreement Study. J Imaging. 2022 Apr 15;8(4):111. doi: 10.3390/jimaging8040111. PMID 35448238